CLINICAL TRIAL: NCT05831020
Title: Method of Securing Skin Graft: A Comparison of Vacuum Assisted Closure Device Versus Bolster Dressing
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dow University of Health Sciences (Other)
Responsible Party: Principal Investigator, Saira Ahmed Chhotani, Dr., Dow University of Health Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB2125/DUHS/Approval/2021/637
Record Dates: First submitted 2023-04-14; First posted 2023-04-26 (Actual); Last update posted 2023-04-26 (Actual); Status verified 2023-04

CONDITIONS: Skin Graft Detachment
Keywords: Graft take, vacuum assisted, Bolster dressing

STUDY DESIGN:
Intervention Model Description: A two arm parallel assignment, where group A will be VAC group and group B will be bolster dressing group.
Who Masked: Outcomes Assessor
Masking Description: The dressing is opened by principal investigator and then the supervising consultant is called for outcome assessment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (VAC group) (Active Comparator): For Group A, VAC dressing was placed to secure split thickness skin graft. Two sheets of sterilized VAC sponge that was cut to fit the wound contour were placed with a fenestrated tube between the two layers that was secured to the surrounding skin using tincture of benzoin spray and an adhesive dressing (OPSITE). The VAC was placed to intermittent -125 mmHg suction for 2 hours and then decompressed for next 2 hours.
  Interventions: Other: VAC and bolster dressing
- Group B (Bolster dressing group) (Active Comparator): For Group B, Bolster dressing was done to secure split thickness skin graft. The recipient site was bolstered with wet bulky cotton gauze dressing and wrapped with cotton bandage. 0.9% normal saline was used for moisture.
  Interventions: Other: VAC and bolster dressing

INTERVENTIONS:
Other: VAC and bolster dressing — Bolster dressing- Moist bulky cotton gauze dressing and wrapped with cotton bandage.
  Vacuum assisted closure (VAC) dressing- A fenestrated tube placed between two sheets of sterilized foam secured to the surrounding skin using adhesive dressing (OPSITE).

SUMMARY:
The goal of this randomized controlled trial is to compare the outcomes of vacuum assisted closure device versus conventional bolster dressing in securing split thickness skin graft in traumatic wounds; with emphasis on percentage of graft take and postoperative complications like hematoma, seroma and infection of graft site. Two groups were formed with 70 patients in each group. Patients were randomly allocated either to group A(VAC group) or group B(bolster dressing group) and outcomes were assessed on 5th post-operative day when first dressing change was done

DETAILED DESCRIPTION:
This randomized controlled trial was conducted at the Department of Plastic and Reconstructive Surgery at Dr. Ruth K.M. Pfau Civil Hospital Karachi from 21st October 2021 to 20th June 2022. Before conducting the study, ethical approval was obtained from Dow University of Health Sciences (DUHS) (IRB-2125/DUHS/Approval/2021/637).

All patients were enrolled via non-probability consecutive sampling. The sample size for the current study was calculated as follows:

Mean graft take for VAC group = 96 ±6 Mean graft take for conventionally treated group = 89±20 (10) Level of confidence = 95% Power = 80% A sample of 140 patients (70 per group) was required to detect mean difference of 7 in graft take between two groups as estimated by using the above parameters through online available calculator Open Epi.

Patients visiting outpatient department and requiring skin graft were admitted to Plastic surgery and recruited into the study with their consent. Study purpose and risk and benefits associated with the procedure were explained to the patient to obtain their consent. Total 70 patients in each group, meeting the inclusion criteria were enrolled. Patients were randomly allocated either to the conventional group or new technique group. Random allocation of patients was done using the SNOSE (sequentially numbered opaque sealed envelope) protocol. Total 140 sequentially numbered opaque sealed envelopes was prepared enclosing the group name with half of the envelop will be enclosing name of group A (VAC group) and other half enclosing the group b (bolster dressing group) and after that envelops was shuffled to ensure randomization.

Skin grafting was performed under general anesthesia. Humby's knife was used to harvest skin graft from donor site. Skin graft was hand meshed and secured to the recipient site circumferentially with absorbable sutures, followed by Tincture of benzoin soaked paraffin gauze layer. For the bolster dressing group, the recipient site was bolstered with wet bulky cotton gauze dressing and wrapped with cotton bandage. 0.9% normal saline was used for moisture. For the Vacuum assisted closure (VAC) Group, two sheets of sterilized VAC sponge that was cut to fit the wound contour were placed with a fenestrated tube between the two layers that was secured to the surrounding skin using tincture of benzoin spray and an adhesive dressing (OPSITE). The VAC was placed at -125mmHg suction and checked for any air leak. Any loss of suction was treated by reinforcing the adhesive dressing over the air leak. The VAC was decompressed and clamped till the patient is shifted back to the ward. Once in ward, The VAC was placed to intermittent -125 mmHg suction for 2 hours and then decompressed for next 2 hours. Bed rest, sling or splint was used for immobilization depending on the location of injury.

Patients were permitted for slight movement for personal hygiene reasons. First dressing change was done on 5th post-operative day. They underwent early change of dressing in case excessive soakage of dressing with blood, serous fluid or foul smelling discharge or pus was present. Dressing of patient was opened on 5th operative day by researcher and then assessed by supervising consultant for percentage of skin graft take and post-operative complications. A pre-designed proforma was designed to collect the data. Patients' data was kept confidential. Medical record no. of patients was tagged with other serial number to assure the confidentiality of the data and only principal investigator had an access to original data.

Data was entered and analyzed by using SPSS version 21. Qualitative variables like gender, socioeconomic status, place of residence, smoking status, medical comorbidities (such as diabetes mellitus and hypertension), graft site, donor site, post-operative complications were presented as frequency with percentages. Quantitative variables such as age, height, weight, BMI, graft size, length of stay in the hospital, percentage of graft take were summarized in terms of mean standard deviation. Effect-modifiers such as age, gender, BMI, smoking status, graft site, graft size, diabetes and hypertension will be controlled through stratification. Post-stratification independent t-test or Mann Whitney U test will be applied to compare percentage of graft take among two treatment groups. Post-stratification chi-square test will be applied to assess difference of post-operative complications among two treatment groups. P-value <0.05 was considered as statistically significant.

ELIGIBILITY:
Inclusion Criteria:

All patients undergoing skin graft at the Civil Hospital

1. aged 18 years to 60 years
2. either gender
3. ASA grade 1
4. Traumatic wounds of size 25 cm2 to 225 cm2 and of greater than 14 days duration with healthy granulation tissue and
5. Consenting to participate in the study.

Exclusion Criteria:

1. Patients with signs of wound infection
2. Patients with wounds of poor blood supply
3. Patients known for allergy or sensitivity to acrylic adhesives.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 140 (Actual)
Dates: Start 2021-10-21 (Actual); Primary Completion 2022-06-20 (Actual); Study Completion 2022-06-20 (Actual)

PRIMARY OUTCOMES:
Graft take | 5th post-operative day or earlier if excessive soakage of dressing
  Defined as the percentage of the skin graft which is adherent to the recipient wound which is wound size. The area for wound size will be pre-operatively measured using ruler in centimeter square and the area where graft is adherent will be measured in percentage. It will be visually assessed by consultant surgeon at the time of first dressing change

SECONDARY OUTCOMES:
Post-operative complications | 5th post-operative day or earlier if excessive soakage of dressing
  Hematoma, seroma and wound infection will be assessed visually by the consultant surgeon on first dressing change.

CONTACTS AND LOCATIONS:
Overall Officials: Saira A Chhotani, MBBS, Principal Investigator — Dow University of Health Sciences
Locations (1):
- Dow University of Health Sciences, Karachi, Pakistan

IPD SHARING:
Plan to Share IPD: No
To maintain confidentiality of participants, medical record no. of patients was tagged with other serial number and only principal investigator had and will have an access to original data.

REFERENCES:
- [Background] Mohsin M, Zargar HR, Wani AH, Zaroo MI, Baba PUF, Bashir SA, Rasool A, Bijli AH. Role of customised negative-pressure wound therapy in the integration of split-thickness skin grafts: A randomised control study. Indian J Plast Surg. 2017 Jan-Apr;50(1):43-49. doi: 10.4103/ijps.IJPS_196_16. PMID 28615809
- [Background] Scherer LA, Shiver S, Chang M, Meredith JW, Owings JT. The vacuum assisted closure device: a method of securing skin grafts and improving graft survival. Arch Surg. 2002 Aug;137(8):930-3; discussion 933-4. doi: 10.1001/archsurg.137.8.930. PMID 12146992
- [Background] Lee SH, Kim YJ. Effectiveness of double tie-over dressing compared with bolster dressing. Arch Plast Surg. 2018 May;45(3):266-270. doi: 10.5999/aps.2017.01424. Epub 2018 May 15. PMID 29788688
- [Background] Dhillon M, Carter CP, Morrison J, Hislop WS, Currie WJ. A comparison of skin graft success in the head & neck with and without the use of a pressure dressing. J Maxillofac Oral Surg. 2015 Jun;14(2):240-2. doi: 10.1007/s12663-014-0618-8. Epub 2014 Feb 11. PMID 26028841
- [Background] Azzopardi EA, Boyce DE, Dickson WA, Azzopardi E, Laing JH, Whitaker IS, Shokrollahi K. Application of topical negative pressure (vacuum-assisted closure) to split-thickness skin grafts: a structured evidence-based review. Ann Plast Surg. 2013 Jan;70(1):23-9. doi: 10.1097/SAP.0b013e31826eab9e. PMID 23249474
- [Background] Kucharzewski M, Mieszczanski P, Wilemska-Kucharzewska K, Taradaj J, Kuropatnicki A, Sliwinski Z. The application of negative pressure wound therapy in the treatment of chronic venous leg ulceration: authors experience. Biomed Res Int. 2014;2014:297230. doi: 10.1155/2014/297230. Epub 2014 Feb 18. PMID 24696847
- [Background] Yadav S, Rawal G, Baxi M. Vacuum assisted closure technique: a short review. Pan Afr Med J. 2017 Nov 21;28:246. doi: 10.11604/pamj.2017.28.246.9606. eCollection 2017. PMID 29881491